CLINICAL TRIAL: NCT04418765
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study With an Extension Period to Evaluate the Efficacy and Safety of Eptinezumab for the Prevention of Migraine in Patients With Unsuccessful Prior Preventive Treatments
Brief Title: A Study to Evaluate the Efficacy and Safety of Eptinezumab for the Prevention of Migraine in Participants That Are Not Helped by Previous Preventive Treatments
Acronym: DELIVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18898A
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo matching to eptinezumab by IV infusion, every 12 weeks starting from Baseline (Day 0) through Week 24.
  Interventions: Drug: Placebo
- Eptinezumab 100 mg (Experimental): Participants will receive eptinezumab 100 mg by IV infusion, every 12 weeks starting from Baseline (Day 0) through Week 24.
  Interventions: Drug: Eptinezumab
- Eptinezumab 300 mg (Experimental): Participants will receive eptinezumab 300 mg by IV infusion, every 12 weeks starting from Baseline (Day 0) through Week 24.
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab, concentrate for solution for infusion 100 mg/milliliter (mL)
  Arms: Eptinezumab 100 mg; Eptinezumab 300 mg
Drug: Placebo — concentrate for solution for infusion, intravenously
  Arms: Placebo

SUMMARY:
Evaluation of eptinezumab in the prevention of migraine in participants with unsuccessful prior preventive treatments.

DETAILED DESCRIPTION:
The total study duration from the screening visit to the completion visit is approximately 76 weeks and includes a screening period (28-30 days), a placebo-controlled treatment period (24 weeks) and a treatment extension period (48 weeks).

The participant will start treatment at the baseline visit and follow a 12-week dosing schedule with either eptinezumab (100 or 300 milligrams [mg]) or placebo by intraveneous (IV) infusion. Participants who were assigned to placebo in the placebo-controlled treatment period, will be randomly allocated to one of two treatment groups: eptinezumab 300 mg or eptinezumab 100 mg.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine, with a history of chronic or episodic migraines of at least 12 months prior to the Screening Visit
* The participant has a migraine onset of ≤50 years of age.
* The participant has ≥4 migraine days per month for each month within the past 3 months prior to the Screening Visit.
* The participant has demonstrated compliance with the Headache eDiary by entry of data for at least 24 of the 28 days following the Screening Visit.
* The participant fulfils the following criteria for chronic migraine (CM) or episodic migraine (EM) in prospectively collected information in the eDiary during the screening period:
* For participants with CM: Migraine occurring on ≥8 days and headache occurring on >14 days
* For participants with EM: Migraine occurring on ≥4 days and headache occurring on ≤14 days
* The participant has documented evidence of treatment failure (must be supported by medical record or by physician's confirmation specific to each treatment) in the past 10 years of 2-4 different migraine preventive medications.
* The participant has a history of either previous or active use of triptans for migraine.

Exclusion Criteria:

* The participant has experienced failure on a previous treatment targeting the calcitonin gene-related peptide (CGRP) pathway.
* The participant has a treatment failure on valproate/divalproex or botulinum toxin A/B and the treatment is not the latest preventive medication prior to study inclusion. The medication is regarded as the latest if the medication start date is after the start date of the other preventive medications and the medication stop date is after the stop date of the other preventive medications.
* The participant has confounding and clinically significant pain syndromes, (for example, fibromyalgia, chronic low back pain, complex regional pain syndrome).
* The participant has a diagnosis of acute or active temporomandibular disorder.
* The participant has a history or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), ophthalmoplegic migraine, and migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration).
* The participant has a psychiatric condition that is uncontrolled and/or untreated for a minimum of 6 months prior to the Screening Visit. Participants with a lifetime history of psychosis and/or mania in the last 5 years prior to the Screening Visit are excluded.
* The participant has a history of clinically significant cardiovascular disease or vascular ischaemia or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).

Other in- and exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (138):
- United States (14):
  - Diablo Clinical Research, Walnut Creek, California
  - Sarkis Clinical Trials - Gainesville, Gainesville, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute Inc. - Minneapolis, Minneapolis, Minnesota
  - Albuqerque Clinical Trials, Albuquerque, New Mexico
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Integrative Clinical Trials, Brooklyn, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Hometown Urgent Care & Occupational Health/Hometown Research - Huber Heights, Dayton, Ohio
  - Lynn Health Science Institute - Oklahoma City, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions - Memphis, Memphis, Tennessee
  - Northwest Clinical Research Center (NWCRC), Bellevue, Washington
  - Northwest Neurological, Spokane, Washington
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Limburg
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment in Neurology and Psychiatry Sveti Naum, Sofia, Sofia-Grad
  - First Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment Heart and Brain EAD, Pleven
  - Medical Center - Teodora EOOD, Rousse
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - Medical Center Medica Plus, Veliko Tarnovo
- Czechia (15):
  - MUDr. Helena Hojdíkova s.r.o. Neurologicka Ambulance, Hradec Králové, Hradec Kralové
  - Vestra Clinics, Rychnov nad Kněžnou, Hradec Kralové
  - CCR Brno, Brno, Jihormoravsky Kraj
  - Fakultni nemocnice Ostrava, Ostrava-Poruba-Poruba, Moravian-Silesian
  - CCR Prague, Prague, Prague
  - Fakultní Thomayerova nemocnice, Prague, Prague
  - Neurologicka Ambulance - Forbeli, Prague, Prague
  - Neuropsychiatrie S.R.O., Prague, Prague
  - Institut Neuropsychiatrické Péce, Prague, Prague
  - CCR Ostrava, Ostrava, Severomoravsky Kraj
  - Fakultní Nemocnice u sv. Anny v Brne, Brno, South Moravian
  - Nemocnice Jihlava, Jihlava
  - Neurosanatio s.r.o, Litomyšl
  - Neurologie, MP-neuro s.r.o., poliklinika Modry pavilon, Slezská Ostrava
  - NeuroMed Zlín s.r.o., Zlín
- Denmark (3):
  - Rigshospitalet Glostrup, Glostrup Municipality, Capital Region
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Sydvestjysk Sygehus - Esbjerg, Esbjerg
- Finland (5):
  - Tampereen Yliopistollinen Sairaala, Tampere, Länsi-Suomen Lääni
  - Terveystalo Ruoholahti, Helsinki, Southern Finland
  - Terveystalo Turku Pulssi, Turku, Western Finland
  - Itä-Suomen Yliopisto - Kuopion Kampus, Kuopio
  - Terveystalo Tampere, Tampere
- France (6):
  - Hôpital Cimiez, Nice, Côte-d'Or
  - Hôpital Charles-Nicolle, Rouen, Haute-Normandie
  - Hôpital Roger Salengro, Lille, Nord
  - Centre Hosptitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Assistance Publique Hôpitaux de Marseille, Marseille, Provence Alpes Cote D'Azure
  - Hôpital Pierre Wertheimer, Bron, Rhone-Alps
- Georgia (10):
  - Helsicore - Israeli-Georgian Medical Research Clinic, Tbilisi, K'alak'i T'bilisi
  - LLC Todua Clinic, Tbilisi, K'alak'i T'bilisi
  - Pineo Medical Ecosystem, Tbilisi
  - Archangel Saint Michael Multiprofile Clinical Hospital, Tbilisi
  - Aversi Clinic - Central Branch, Tbilisi
  - Mediclub Georgia Medical, Tbilisi
  - Jerarsi Clinic, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Center, Tbilisi
  - Simon Khechinashvili University Hospital, Tbilisi
  - Consilium Medulla Multiprofile Clinic, Tbilisi
- Germany (15):
  - Neuroplus, Mannheim, Baden-Wurttemberg
  - MVZ Dr. Roth & Kollegen GbR, Ostfildern, Baden-Wurttemberg
  - NeuroConcept AG, Stuttgart, Baden-Wurttemberg
  - Praxis Dr. Steinwachs, Nuremberg, Bavaria
  - CTC North, Hamburg, Hamburg (Hansestadt)
  - Synexus - Prüfzentrum Frankfurt/Main, Frankfurt am Main, Hesse
  - Migräne- und Kopfschmerzklinik Königstein, Königstein im Taunus, Hesse
  - Studienzentrum Nord West, Westerstede, Lower Saxony
  - Neurozentrum Bielefeld, Bielefeld, North Rhine-Westphalia
  - Neurologische Praxis Dr. Stude, Bochum, North Rhine-Westphalia
  - Praxis Astrid Gendolla, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Synexus - Leipzig, Leipzig, Saxony
  - Synexus Clinical Research - Berlin, Berlin
  - Neuropraxis München Süd, Unterhaching
- Hungary (3):
  - Valeomed Diagnosztikai Kozpont, Esztergom, Komarom-Esztergom County
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa, Pest County
  - UNO Medical Trials Kft., Budapest
- Italy (6):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - San Raffaele Pisana, Rome, Roma
  - Universita Campus Bio-Medico di Roma, Roma, Rome
  - Azienda Ospedaliera - Universitaria Sant' Andrea, Roma, Rome
  - IRCCS Istituto Delle Scienze Neurologiche di Bologna, Bologna
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione Mondino - Istituto Neurologico Nazionale a Carattere Scientifico IRCCS, Pavia
- Poland (19):
  - Centrum Medyczne Solumed, Poznan, Greater Poland Voivodeship
  - Synexus - Poznan, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Pratia - Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia dr Boczarska-Jedynak, Oświęcim, Lesser Poland Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - Prywatny Gabinet Lekarski Urszula Chyrchel-Paszkiewicz, Lublin, Lublin Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. n. med. Anna Szczepanska-Szerej, Lublin, Lublin Voivodeship
  - Concept Medica Trials Prywatny Gabinet Lekarski Urszula Chyrchel-Paszkiewicz, Warsaw, Masovian Voivodeship
  - SOMED CR - Warsaw, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by Pratia, Warsaw, Masovian Voivodeship
  - Synexus - Gdynia, Gdynia, Pomeranian Voivodeship
  - Synexus - Czestochowa, Częstochowa, Silesian Voivodeship
  - Synexus - Katowice, Katowice, Silesian Voivodeship
  - Neuro-Care Katowice, Siemianowice Śląskie, Silesian Voivodeship
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag, Warmian-Masurian Voivodeship
  - Centrum Medyczne Pratia - Czestochowa, Częstochowa
  - SOMED CR - Lodz, Lodz
- University Headache Clinic, Moscow, Russia
- Slovakia (4):
  - Neurologicka ambulancia MUDr. Dupejova s.r.o., Banská Bystrica
  - In Medic, Bardejov
  - MEDBAJ s.r.o., Dolný Kubín
  - Medicínske Centrum Konzílium - Dubnica nad Vahom, Dubnica nad Váhom
- Spain (11):
  - Hospital Universitario de Basurto, Bilbao, Biscay
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital Alvaro Cunqueiro - Clinico Universitario Vigo, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Sweden (4):
  - Migränkliniken Europa AB, Värnamo, Kronoborgs Län
  - Stortorgets neurologmottagning, Helsingborg, Skåne County
  - Centralsjukhuset Kristianstad, Kristianstad, Skåne County
  - Universitetssjukhuset i Linköping, Linköping, Östergötland County
- United Kingdom (12):
  - Synexus - Scotland Clinical Research Centre, Bellshill, England
  - Synexus - The Lancashire Clinic, Chorley, England
  - Synexus Midlands Clinical Research Centre, Edgbaston, England
  - Synexus - The Hexham Clinic, Hexham, England
  - Synexus - Merseyside Clinical Research Centre, Liverpool, England
  - Panthera Biopartners - North London, London, England
  - Synexus - Manchester Clinical Research Centre, Manchester, England
  - Panthera Biopartners - Manchester, Manchester, England
  - Panthera Biopartners - Preston, Preston, England
  - Synexus - Thames Valley Clinical Research Centre, Reading, England
  - Northern Care Alliance NHS Foundation Trust, Salford, England
  - Synexus - Wales, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pozo-Rosich P, Tassorelli C, Boserup LP, Awad SF, Lee XY, Ailani J. Sustained Efficacy of Eptinezumab in Participants with Migraine for Whom Prior Preventive Treatments Failed and Who Self-reported Psychiatric Comorbidities: Post Hoc Analysis of the Placebo-controlled DELIVER Trial. Neurol Ther. 2026 Feb 11. doi: 10.1007/s40120-026-00893-4. Online ahead of print. PMID 41670910
- [Derived] Tassorelli C, Starling AJ, Awad SF, Lee XY, Boserup LP, Asher D, Soni-Brahmbhatt S, Sperling B, Goadsby PJ. Early and Sustained Shift in Headache Day Frequency Following Eptinezumab Treatment in Adults With Migraine for Whom 2-4 Previous Preventive Treatments Have Failed: A Post Hoc Analysis of the Randomized DELIVER Trial. Eur J Neurol. 2025 Dec;32(12):e70460. doi: 10.1111/ene.70460. PMID 41395928
- [Derived] Barbanti P, Awad SF, Rae-Espinoza H, Regnier SA, Lee XY, Goadsby PJ. Impact of eptinezumab on work productivity beyond reductions in monthly migraine days: post hoc analysis of the DELIVER trial. J Patient Rep Outcomes. 2024 Dec 18;8(1):146. doi: 10.1186/s41687-024-00813-w. PMID 39692817
- [Derived] Jonsson L, Awad SF, Regnier SA, Talon B, Kymes S, Lee XY, Goadsby PJ. Structural equation modeling for identifying the drivers of health-related quality of life improvement experienced by patients with migraine receiving eptinezumab. J Headache Pain. 2024 Mar 28;25(1):45. doi: 10.1186/s10194-024-01752-z. PMID 38549121
- [Derived] Pozo-Rosich P, Ashina M, Tepper SJ, Jensen S, Boserup LP, Josiassen MK, Sperling B. Eptinezumab Demonstrated Efficacy Regardless of Prior Preventive Migraine Treatment Failure Type: Post Hoc Analyses of the DELIVER Study. Neurol Ther. 2024 Apr;13(2):339-353. doi: 10.1007/s40120-023-00575-5. Epub 2024 Jan 18. PMID 38236314
- [Derived] Ashina M, Tepper SJ, Gendolla A, Sperling B, Ettrup A, Josiassen MK, Starling AJ. Long-term effectiveness of eptinezumab in patients with migraine and prior preventive treatment failures: extension of a randomized controlled trial. J Headache Pain. 2023 Nov 20;24(1):155. doi: 10.1186/s10194-023-01688-w. PMID 37985968
- [Derived] Jonsson L, Regnier SA, Kymes S, Awad SF, Talon B, Lee XY, Goadsby PJ. Estimating treatment effects on health utility scores for patients living with migraine: a post hoc analysis of the DELIVER trial. Expert Rev Pharmacoecon Outcomes Res. 2023 Jul-Dec;23(7):797-803. doi: 10.1080/14737167.2023.2219898. Epub 2023 Jun 2. PMID 37256558
- [Derived] Ashina M, Lanteri-Minet M, Ettrup A, Christoffersen CL, Josiassen MK, Phul R, Sperling B, Pozo-Rosich P. Efficacy and safety of eptinezumab for migraine prevention in patients with prior preventive treatment failures: subgroup analysis of the randomized, placebo-controlled DELIVER study. Cephalalgia. 2023 May;43(5):3331024231170807. doi: 10.1177/03331024231170807. PMID 37125484
- [Derived] Goadsby PJ, Barbanti P, Lambru G, Ettrup A, Christoffersen CL, Josiassen MK, Phul R, Sperling B. Eptinezumab improved patient-reported outcomes and quality of life in patients with migraine and prior preventive treatment failures. Eur J Neurol. 2023 Apr;30(4):1089-1098. doi: 10.1111/ene.15670. Epub 2023 Jan 21. PMID 36583633
- [Derived] Barbanti P, Goadsby PJ, Lambru G, Ettrup A, Christoffersen CL, Josiassen MK, Phul R, Sperling B. Effects of eptinezumab on self-reported work productivity in adults with migraine and prior preventive treatment failure in the randomized, double-blind, placebo-controlled DELIVER study. J Headache Pain. 2022 Dec 2;23(1):153. doi: 10.1186/s10194-022-01521-w. PMID 36460983
- [Derived] Ashina M, Lanteri-Minet M, Pozo-Rosich P, Ettrup A, Christoffersen CL, Josiassen MK, Phul R, Sperling B. Safety and efficacy of eptinezumab for migraine prevention in patients with two-to-four previous preventive treatment failures (DELIVER): a multi-arm, randomised, double-blind, placebo-controlled, phase 3b trial. Lancet Neurol. 2022 Jul;21(7):597-607. doi: 10.1016/S1474-4422(22)00185-5. PMID 35716692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 2 periods: Placebo-controlled Period - 24-week double-blind treatment period with placebo or eptinezumab and Extension Period - 48-week dose-blinded period with eptinezumab after completion of the Placebo-controlled Period.
Pre-assignment Details: Participants assigned to placebo in the Placebo-controlled Period were randomized 1:1 to treatment with either eptinezumab 100 milligrams (mg) or eptinezumab 300 mg. Participants assigned to eptinezumab 100 mg or 300 mg in the Placebo-controlled Period continued their treatment.
Groups:
- Placebo: Participants received placebo matched to eptinezumab by intravenous (IV) infusion on Baseline (Day 0) and on Week 12 in the double-blind treatment period.
- Eptinezumab 100 mg: Participants received eptinezumab 100 mg by IV infusion on Baseline (Day 0); and thereafter, every 12 weeks up to Week 60 (2 doses in the double-blind treatment period and 4 doses in the dose-blinded extension period).
- Eptinezumab 300 mg: Participants received eptinezumab 300 mg by IV infusion on Baseline (Day 0); and thereafter, every 12 weeks up to Week 60 (2 doses in the double-blind treatment period and 4 doses in the dose-blinded extension period).
Period: Placebo-controlled Period (24 Weeks)
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Started | 299 | 299 | 294
Received at Least 1 Dose of Study Drug | 298 | 299 | 294
Completed | 293 | 288 | 284
Not Completed | 6 | 11 | 10
Not completed — Adverse Event | 1 | 1 | 6
Not completed — Lack of Efficacy | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other than specified | 2 | 0 | 1
Not completed — Randomized but not treated | 1 | 0 | 0
Period: Extension Period (48 Weeks)
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Started | 0 | 433 (145 participants assigned to placebo in the Placebo-controlled Period were randomized to eptinezumab 100 mg.) | 432 (148 participants assigned to placebo in the Placebo-controlled Period were randomized to eptinezumab 300 mg.)
Received at Least 1 Dose of Study Drug | 0 | 433 | 432
Completed | 0 | 392 | 390
Not Completed | 0 | 41 | 42
Not completed — Adverse Event | 0 | 2 | 9
Not completed — Lack of Efficacy | 0 | 13 | 13
Not completed — Withdrawal by Subject | 0 | 21 | 14
Not completed — Non-compliance with study drug | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Other than specified | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who had a valid baseline assessment and at least 1 valid post-baseline 4-week assessment of monthly migraine days (MMDs) in Weeks 1 to 12.
Groups:
- Placebo: Participants received placebo matched to eptinezumab by IV infusion on Baseline (Day 0) and on Week 12 in the double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg | Total
Number analyzed (Participants) | 298 | 299 | 293 | 890
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.83) | 44.6 (10.76) | 43.1 (10.2) | 43.8 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 277 | 260 | 800
  Male | 35 | 22 | 33 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 285 | 288 | 281 | 854
  Race: Other | 2 | 0 | 0 | 2
  Race: Unknown | 11 | 11 | 12 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 1 | 1
  Ethnicity: Not Hispanic or Latino | 2 | 1 | 2 | 5
  Ethnicity: Not collected | 296 | 298 | 290 | 884
Monthly Migraine Days (MMDs) [Mean (Standard Deviation); unit: days/month] — A migraine day was defined as any day the participant reported a headache that met criterion A, B, C, or D as defined in the outcome measure 1.
  days/month | 13.9 (5.72) | 13.8 (5.58) | 13.7 (5.44) | 13.8 (5.57)
Monthly Headache Days (MHDs) [Mean (Standard Deviation); unit: days/month] — A headache day was defined as a day with a headache that lasted ≥30 minutes or met the definition of a migraine day (as defined in criterion A, B, C, or D in outcome measure 1).
  days/month | 14.5 (5.79) | 14.5 (5.63) | 14.4 (5.45) | 14.5 (5.62)
Headache Impact Test (HIT-6) Score [Mean (Standard Deviation); unit: units on a scale] — HIT-6 (version 1.0) is a Likert-type, self-reporting questionnaire designed to assess the impact of an occurring headache and its effect on the ability to function normally in daily life. The HIT-6 contains 6 questions, each item was rated from never to always with the following response scores: never = 6, rarely = 8, sometimes = 10, very often = 11, and always = 13. The total score for the HIT-6 was the sum of each response score ranging from 36 to 78. The life impact derived from the total score was described as followed: severe (≥60), substantial (56-59), some (50-55), little to none (≤49). Population: Here, number analyzed = participants evaluable for this baseline measure.
  units on a scale
    number analyzed (Participants) | 288 | 281 | 287 | 856
    (all) | 66.2 (4.38) | 66.6 (4.7) | 66.5 (4.41) | 66.4 (4.5)
Percentage of Migraine Attacks With Severe Pain Intensity [Mean (Standard Deviation); unit: percentage of migraine attacks] — A migraine attack was defined as a headache that occurred on a single day or lasted >1 day and that met the criteria for a migraine day (as defined in criterion A, B, C, or D in outcome measure 1).
  percentage of migraine attacks | 40.4 (29.74) | 47.1 (29.82) | 43.9 (28.4) | 43.8 (29.43)
Percentage of Headache Episodes With Severe Pain Intensity [Mean (Standard Deviation); unit: percentage of headache episodes] — A headache episode was defined as a headache lasted ≥30 minutes or that met the criteria for a migraine (as defined in criterion A, B, C, or D in outcome measure 1).
  percentage of headache episodes | 38.5 (29.29) | 44.2 (28.56) | 41 (27.01) | 41.2 (28.38)
Acute Migraine Medication Days [Mean (Standard Deviation); unit: days] — Population: Here, number analyzed = participants evaluable for this baseline measure.
  days
    number analyzed (Participants) | 298 | 299 | 292 | 889
    (all) | 11.2 (5.93) | 11.2 (5.47) | 11 (5.29) | 11.1 (5.57)
MMDs With Use of Acute Medication [Mean (Standard Deviation); unit: days/month] | 12.5 (5.62) | 12.7 (5.48) | 12.4 (5.38) | 12.5 (5.49)
Migraine-Specific Quality of Life (MSQ) Subscores [Mean (Standard Deviation); unit: units on a scale] — The MSQ is a participant-reported outcome designed to assess the quality of life in participants with migraine. It consists of 14 items covering 3 domains: role function restrictive (7 items); role function preventive (4 items); and emotional function (3 items). Each item was scored on a 6-point scale ranging from 1 (none of the time) to 6 (all of the time). Raw domain scores were summed and transformed to a 0- to 100-point scale. Higher scores indicated better quality of life. Population: Here, number analyzed = participants evaluable for this baseline measure.
  units on a scale
    MSQ role function-restrictive: number analyzed (Participants) | 288 | 276 | 287 | 851
    MSQ role function-restrictive | 35.1 (17.14) | 35.7 (17.33) | 35.7 (16.68) | 35.5 (17.03)
    MSQ role function-preventive: number analyzed (Participants) | 288 | 276 | 287 | 851
    MSQ role function-preventive | 50.5 (22.14) | 50.2 (21.39) | 51 (21.47) | 50.6 (21.65)
    MSQ emotional function: number analyzed (Participants) | 288 | 276 | 287 | 851
    MSQ emotional function | 48.4 (26.63) | 50.3 (24.7) | 48.6 (23.8) | 49.1 (25.06)
Health-Related Quality of Life (EQ-5D-5L) Visual Analog Scale (VAS) Score [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D-5L is a participant-reported assessment designed to measure the participant's well-being. It consists of 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a VAS of the overall health state. Each descriptive item was rated on a 5-point index ranging from 1 (no problems) to 5 (extreme problems). The VAS ranged from 0 (worst imaginable health state) to 100 (best imaginable health state). Population: Here, number analyzed = participants evaluable for this baseline measure.
  units on a scale
    number analyzed (Participants) | 287 | 276 | 285 | 848
    (all) | 74 (20.36) | 75.9 (19.01) | 74.5 (20.72) | 74.8 (20.05)
WPAI Questionnaire Subscores (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment [Mean (Standard Deviation); unit: units on a scale] — WPAI Questionnaire contains 6 items that measure: 1) employment status, 2) hours missed from work due to specific health problem, 3) hours missed from work for other reasons, 4) hours actually worked, 5) degree health affected productivity while working, and 6) degree health affected productivity in regular unpaid activities. Four scores were calculated from the responses to these 6 items: absenteeism, presenteeism, work productivity loss, and activity impairment. Scores were calculated as impairment percentages (0-100%), with higher numbers indicating greater impairment and less productivity. Population: Here, number analyzed = participants evaluable for this baseline measure.
  units on a scale
    WPAI Absenteeism: number analyzed (Participants) | 218 | 196 | 209 | 623
    WPAI Absenteeism | 12.8 (20.7) | 11.4 (19.4) | 12 (19.31) | 12.1 (19.58)
    WPAI Presenteeism: number analyzed (Participants) | 212 | 191 | 206 | 609
    WPAI Presenteeism | 51.7 (24.22) | 50.8 (25.61) | 53.3 (24.01) | 52 (24.58)
    WPAI Work productivity loss: number analyzed (Participants) | 212 | 191 | 206 | 609
    WPAI Work productivity loss | 55.6 (24.7) | 53.7 (26.17) | 57 (24.1) | 55.5 (24.97)
    WPAI Activity impairment: number analyzed (Participants) | 286 | 274 | 285 | 845
    WPAI Activity impairment | 58.7 (23.52) | 58.5 (23.47) | 59.1 (23.37) | 58.7 (23.43)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Monthly Migraine Days (MMDs) Averaged Over Weeks 1 to 12
Description: A migraine day was defined as any day the participant reported a headache that met criterion A, B, C, or D: Criterion A (all of the following criteria): lasted ≥4 hours, had ≥2 of the following: unilateral location; pulsating quality; moderate or severe pain intensity; aggravation by, or causing avoidance of, routine physical activity; and was accompanied by ≥1 of the following: nausea; vomiting; photophobia and phonophobia. Criterion B: lasted ≥30 minutes and the participant had an aura with the headache. Criterion C: lasted ≥30 minutes and met ≥2 of the following criteria: lasted ≥4 hours, had ≥2 of the following: unilateral location; pulsating quality; moderate or severe pain intensity; aggravation by, or causing avoidance of, routine physical activity, and was accompanied by ≥1 of the following: nausea; vomiting; photophobia and phonophobia. Criterion D: the participant took medication to treat the headache because he/she believed he/she was having a migraine.
Time Frame: Baseline, Weeks 1 - 12
Population: FAS included all randomized participants who had a valid baseline assessment and at least 1 valid post-baseline 4-week assessment of MMDs in Weeks 1 to 12.
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
days/month | -2.1 (0.38) | -4.8 (0.37) | -5.3 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Eptinezumab 300 mg; Analysis was performed using a restricted maximum likelihood (REML)-based mixed model for repeated measurements (MMRM) with month (Weeks 1-4, 5-8, 9-12, 13-16, 17-20, 21-24), country, stratification factor (monthly MHDs at baseline: ≤14/>14) and treatment as factors, baseline score as a continuous covariate, treatment-by-month interaction, baseline score-by-month interaction, and stratum-by-month interaction. A testing strategy was applied to ensure protection of the type 1 error; Test type: Other — Testing sequence: 1. Change in MMDs (Weeks 1-12) 300 mg vs placebo; 2. 50% responders for MMDs (Weeks 1-12) 300 mg vs placebo; 3. Change in MMDs (Weeks 1-12) 100 mg vs placebo; 4. 50% responders for MMDs (Weeks 1-12) 100 mg vs placebo; 5a. Change in MMDs (Weeks 13-24), 5b. 75% responders for MMDs (Weeks 1-12), 5c. Change in HIT-6 (Week 12) 300 mg vs placebo; 6a. Change in MMDs (Weeks 13-24), 6b. 75% responders for MMDs (Weeks 1-12), 6c. Change in HIT-6 (Week 12) 100 mg vs placebo; p < 0.0001, Mixed Models Analysis — Testing continued only, if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 1 of testing order; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-3.9 to -2.5], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo vs Eptinezumab 100 mg; Analysis was performed using an REML-based MMRM with month (Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20, Weeks 21-24), country, stratification factor (monthly MHDs at baseline: ≤14/>14) and treatment as factors, baseline score as a continuous covariate, treatment-by-month interaction, baseline score-by-month interaction, and stratum-by-month interaction. A testing strategy (sequence of tests) was applied to ensure protection of the type 1 error; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Testing continued only, if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 3 of testing order; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-3.4 to -2.0], Standard Error of Mean 0.36

2. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in MMDs Averaged Over Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline to Weeks 1 - 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 13.1 | 42.1 | 49.5
Statistical Analysis 1: Comparison: Placebo vs Eptinezumab 300 mg; Analysis was performed using logistic regression model including baseline MMDs as a continuous covariate, and treatment and stratification factor (MHD at baseline: ≤14/>14) as factors. A testing strategy (sequence of tests) was applied to ensure protection of the type 1 error; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic — Testing continued only, if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 2 of testing order; Odds Ratio (OR) = 6.58, 95% CI 2-sided [4.41 to 10.01]
Statistical Analysis 2: Comparison: Placebo vs Eptinezumab 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic — Testing continued only, if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 4 of testing order; Odds Ratio (OR) = 4.91, 95% CI 2-sided [3.29 to 7.47]

3. Secondary Outcome: Change From Baseline in the Number of MMDs Averaged Over Weeks 13 to 24
Description: as for outcome 1
Time Frame: Baseline, Weeks 13 - 24
Population: FAS included all randomized participants who had a valid baseline assessment and at least 1 valid post-baseline 4-week assessment of MMDs in Weeks 1 to 12. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 295 | 287 | 286
days/month | -2.4 (0.39) | -5.4 (0.39) | -6.1 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Eptinezumab 300 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 5a of testing order; Testing continued only, if the previous comparison was statistically significant; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-4.5 to -3.0], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Placebo vs Eptinezumab 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Threshold for significance: The consecutive order of the smallest (p1), the second smallest (p2), and the largest p-value (p3) had to be <α/3, <α/2, and <α, where α = 0.05. Here it is test no. 6a of testing order; Testing continued only, if the previous comparison was statistically significant; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-3.8 to -2.2], Standard Error of Mean 0.39

4. Secondary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in MMDs Averaged Over Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline to Weeks 1 - 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 2.0 | 15.7 | 18.8
Statistical Analysis 1: Comparison: Placebo vs Eptinezumab 300 mg; Analysis was performed using logistic regression model including baseline MMDs as a continuous covariate, and treatment and stratification factor (MHD at baseline: ≤14/>14) as factors. A testing strategy (sequence of tests) was applied to ensure protection of the type 1 error. Testing continued only, if the previous comparison was statistically significant; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic — Threshold for significance: The consecutive order of the smallest (p1), the second smallest (p2), and the largest p-value (p3) had to be <α/3, <α/2, and <α, where α = 0.05. Here it is test no. 5b of testing order; Odds Ratio (OR) = 11.43, 95% CI 2-sided [5.22 to 30.15]
Statistical Analysis 2: Comparison: Placebo vs Eptinezumab 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic — Threshold for significance: The consecutive order of the smallest (p1), the second smallest (p2), and the largest p-value (p3) had to be <α/3, <α/2, and <α, where α = 0.05. Here it is test no. 6b of testing order; Odds Ratio (OR) = 9.19, 95% CI 2-sided [4.16 to 24.35]

5. Secondary Outcome: Change From Baseline in the Headache Impact Test (HIT-6) Score at Week 12
Description: The HIT-6 (version 1.0) is a Likert-type, self-reporting questionnaire designed to assess the impact of an occurring headache and its effect on the ability to function normally in daily life. The HIT-6 contains 6 questions, each item was rated from never to always with the following response scores: never = 6, rarely = 8, sometimes = 10, very often = 11, and always = 13. The total score for the HIT-6 was the sum of each response score ranging from 36 to 78. The life impact derived from the total score was described as followed: severe (≥60), substantial (56-59), some (50-55), little to none (≤49).
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 288 | 277 | 283
units on a scale | -3.1 (0.61) | -6.9 (0.61) | -8.5 (0.60)
Statistical Analysis 1: Comparison: Placebo vs Eptinezumab 300 mg; Analysis was performed using MMRM with the following fixed effects: visit, country, stratification factor (MHDs at baseline: ≤14/>14) and treatment as factors, baseline HIT-6 Total Score as a continuous covariate, baseline score-by-visit interaction, treatment-by-visit interaction, and stratum-by-visit interaction. A testing strategy (sequence of tests) was applied to ensure protection of the type 1 error. Testing continued only, if the previous comparison was statistically significant; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Threshold for significance: The consecutive order of the smallest (p1), the second smallest (p2), and the largest p-value (p3) had to be <α/3, <α/2, and <α, where α = 0.05. Here it is test no. 5c of testing order; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-6.7 to -4.2], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo vs Eptinezumab 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Threshold for significance: The consecutive order of the smallest (p1), the second smallest (p2), and the largest p-value (p3) had to be <α/3, <α/2, and <α, where α = 0.05. Here it is test no. 6c of testing order; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-5.0 to -2.5], Standard Error of Mean 0.63

6. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in MMDs Averaged Over Weeks 13 to 24
Description: as for outcome 1
Time Frame: Baseline to Weeks 13 - 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 295 | 287 | 286
percentage of participants | 23.7 | 52.3 | 59.1

7. Secondary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in MMDs Averaged Over Weeks 13 to 24
Description: as for outcome 1
Time Frame: Baseline to Weeks 13 - 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 295 | 287 | 293
percentage of participants | 6.8 | 21.3 | 27.6

8. Secondary Outcome: Percentage of Participants With 100% Reduction From Baseline in MMDs Averaged Over Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline to Weeks 1 - 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 1.1 | 5.9 | 7.7

9. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in Monthly Headache Days (MHDs) Averaged Over Weeks 1 to 12
Description: A headache day was defined as a day with a headache that lasted ≥30 minutes or met the definition of a migraine day (as defined in criterion A, B, C, or D above in outcome measure 1).
Time Frame: Baseline to Weeks 1 - 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 12.8 | 39.5 | 45.7

10. Secondary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in Monthly Headache Days (MHDs) Averaged Over Weeks 1 to 12
Description: as for outcome 9
Time Frame: Baseline to Weeks 1 - 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 2.3 | 15.1 | 16.4

11. Secondary Outcome: Percentage of Participants With 100% Reduction From Baseline in Monthly Headache Days (MHDs) Averaged Over Weeks 1 to 12
Description: as for outcome 9
Time Frame: Baseline to Weeks 1 - 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 1.1 | 4.1 | 5.3

12. Secondary Outcome: Change From Baseline in the Number of MHDs Averaged Over Weeks 1 to 12
Description: as for outcome 9
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
days/month | -2.1 (0.38) | -4.6 (0.37) | -5.1 (0.37)

13. Secondary Outcome: Change From Baseline in the Percentage of Migraine Attacks With Severe Pain Intensity Averaged Over Weeks 1 to 12
Description: A migraine attack was defined as a headache that occurred on a single day or lasted >1 day and that met the criteria for a migraine day (as defined in criterion A, B, C, or D above in outcome measure 1).
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of migraine attacks
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of migraine attacks | -10.2 (1.91) | -17.9 (1.87) | -21.3 (1.87)

14. Secondary Outcome: Change From Baseline in the Percentage of Headache Episodes With Severe Pain Intensity Averaged Over Weeks 1 to 12
Description: A headache episode was defined as a headache lasted ≥30 minutes or that met the criteria for a migraine (as defined in criterion A, B, C, or D above in outcome measure 1).
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of headache episodes
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of headache episodes | -8.8 (1.85) | -16.2 (1.81) | -19.5 (1.81)

15. Secondary Outcome: Change From Baseline in the Number of Monthly Days With Use of Acute Migraine Medication Averaged Over Weeks 1 to 12
Description: In the evening eDiary, participants were asked each day to fill out whether they used any of the following medications during that day: Ergotamine, triptan, analgesic, opioid, or combination analgesic. A day where the participant answered that they took any of those in the evening eDiary was considered a day with use of acute migraine medication.
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 298 | 290
days/month | -1.6 (0.34) | -4.1 (0.33) | -4.6 (0.34)

16. Secondary Outcome: Change From Baseline in the Number of Monthly Days With Use of Acute Migraine Medication Averaged Over Weeks 13 to 24
Description: as for outcome 15
Time Frame: Baseline, Weeks 13- 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 294 | 287 | 285
days/month | -1.7 (0.36) | -4.6 (0.36) | -5.2 (0.36)

17. Secondary Outcome: Change From Baseline in the Number of MMDs With Use of Acute Medication Averaged Over Weeks 1 to 12
Description: Number of MMDs with acute medication usage was derived using the answer to "Did you take any medications to treat this headache?" in the headache diary. The question was asked when a participant was ending a headache. Thus, a migraine day with acute medication usage was defined as a migraine day with the extra condition that this question was answered as "Yes".
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
days/month | -2.0 (0.36) | -4.6 (0.36) | -5.2 (0.36)

18. Secondary Outcome: Change From Baseline in the Number of MMDs With Use of Acute Medication Averaged Over Weeks 13 to 24
Description: as for outcome 17
Time Frame: Baseline, Weeks 13 - 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 295 | 287 | 286
days/month | -2.1 (0.39) | -4.9 (0.39) | -5.8 (0.38)

19. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Week 12
Description: The PGIC is a single, participant-reported item reflecting the participant's impression of change in his/her disease status since the start of the study (that is, in relation to activity limitations, symptoms, emotions, and overall quality of life). Participants rated their impression of change in disease status on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) where a higher score indicated worsening. Score ranges from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status.
Time Frame: Week 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 297 | 292 | 289
units on a scale | 3.6 (0.09) | 2.6 (0.09) | 2.5 (0.09)

20. Secondary Outcome: PGIC Score at Week 24
Description: as for outcome 19
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 286 | 280 | 281
units on a scale | 3.5 (0.09) | 2.5 (0.09) | 2.4 (0.09)

21. Secondary Outcome: Change From Baseline in the Number of MMDs in Participants With Medication Overuse Headache (MOH) Averaged Over Weeks 1 to 12
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 37 | 38 | 35
days/month | -2.3 (1.12) | -5.6 (1.07) | -7.3 (1.18)

22. Secondary Outcome: Percentage of Participants With Migraine on the Day After First Dosing
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 298 | 299 | 293
percentage of participants | 43.7 | 27.2 | 24.4

23. Secondary Outcome: Most Bothersome Symptom (MBS) Score at Week 12
Description: Participants were asked about their most bothersome symptom associated with their migraines during the Baseline Visit. Participants were asked to rate the improvement in this symptom from baseline on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) where a high score indicated worsening. Score ranges from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status. The MBS areas included: nausea, vomiting, sensitivity to light, sensitivity to sound, mental cloudiness, fatigue, pain with activity, mood changes, and other symptoms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 293 | 289 | 287
units on a scale | 3.7 (0.09) | 2.8 (0.09) | 2.7 (0.09)

24. Secondary Outcome: Change From Baseline in the HIT-6 Score at Week 24
Description: as for outcome 5
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 278 | 266 | 276
units on a scale | -3.9 (0.63) | -8.9 (0.63) | -9.9 (0.62)

25. Secondary Outcome: Change From Baseline in the Migraine-Specific Quality of Life (MSQ) Subscores (Role Function-Restrictive, Role Function-Preventive, Emotional Function) at Week 12
Description: The MSQ is a participant-reported outcome designed to assess the quality of life in participants with migraine. It consists of 14 items covering 3 domains: role function restrictive (7 items); role function preventive (4 items); and emotional function (3 items). Each item was scored on a 6-point scale ranging from 1 (none of the time) to 6 (all of the time). Raw domain scores were summed and transformed to a 0- to 100-point scale. Higher scores indicated better quality of life.
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 288 | 271 | 283
units on a scale
  MSQ Role Function-Restrictive | 13.7 (1.75) | 25.0 (1.75) | 28.7 (1.72)
  MSQ Role Function-Preventive | 11.6 (1.63) | 22.7 (1.64) | 25.0 (1.61)
  MSQ Emotional Function | 9.6 (1.83) | 20.6 (1.84) | 23.1 (1.80)

26. Secondary Outcome: Change From Baseline in the Health-Related Quality of Life (EQ-5D-5L) Visual Analog Scale (VAS) Score at Week 12
Description: The EQ-5D-5L is a participant-reported assessment designed to measure the participant's well-being. It consists of 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a VAS of the overall health state. Each descriptive item was rated on a 5-point index ranging from 1 (no problems) to 5 (extreme problems). The VAS ranged from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 287 | 271 | 281
units on a scale | -3.1 (1.39) | 2.0 (1.40) | 4.4 (1.38)

27. Secondary Outcome: Change From Baseline in the MSQ Subscores (Role Function-Restrictive, Role Function-Preventive, Emotional Function) at Week 24
Description: as for outcome 25
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 278 | 259 | 275
units on a scale
  MSQ Role Function-Restrictive | 15.0 (1.76) | 30.1 (1.78) | 30.0 (1.73)
  MSQ Role Function-Preventive | 13.1 (1.63) | 25.7 (1.65) | 26.3 (1.61)
  MSQ Emotional Function | 9.9 (1.84) | 24.1 (1.86) | 24.1 (1.81)

28. Secondary Outcome: Change From Baseline in the Health-Related Quality of Life (EQ-5D-5L) VAS Score at Week 24
Description: as for outcome 26
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 276 | 258 | 273
units on a scale | -2.8 (1.38) | 2.0 (1.40) | 5.2 (1.37)

29. Secondary Outcome: Change From Baseline in the Work Productivity and Activity Impairment (WPAI) Questionnaire Subscores (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) at Week 12
Description: The WPAI Questionnaire is a participant-reported instrument developed to measure the impact on work productivity and regular activities attributable to a specific health problem (migraine). Recall period is the past 7 days. It contains 6 items that measure: 1) employment status, 2) hours missed from work due to the specific health problem, 3) hours missed from work for other reasons, 4) hours actually worked, 5) degree health affected productivity while working, and 6) degree health affected productivity in regular unpaid activities. Four scores were calculated from the responses to these 6 items: absenteeism, presenteeism, work productivity loss, and activity impairment. Scores were calculated as impairment percentages (0-100%), with higher numbers indicating greater impairment and less productivity, i.e, worse outcomes.
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants who had a valid baseline assessment and at least 1 valid post-baseline 4-week assessment of MMDs in Weeks 1 to 12. Here, overall number of participants analyzed = participants evaluable for this outcome measure. Number analyzed = participants evaluable for specified categories.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 286 | 268 | 280
units on a scale
  Absenteeism: number analyzed (Participants) | 196 | 174 | 183
  Absenteeism | -0.1 (1.49) | -5.8 (1.53) | -3.8 (1.50)
  Presenteeism: number analyzed (Participants) | 188 | 169 | 179
  Presenteeism | -9.9 (2.42) | -19.0 (2.46) | -23.3 (2.40)
  Work productivity loss: number analyzed (Participants) | 188 | 169 | 179
  Work productivity loss | -9.7 (2.56) | -19.5 (2.61) | -24.0 (2.54)
  Activity impairment | -11.2 (2.07) | -21.3 (2.07) | -23.8 (2.05)

30. Secondary Outcome: Change From Baseline in the WPAI Questionnaire Subscores (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) at Week 24
Description: as for outcome 29
Time Frame: Baseline, Week 24
Population: as for outcome 29
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 275 | 256 | 273
units on a scale
  Absenteeism: number analyzed (Participants) | 180 | 151 | 168
  Absenteeism | -0.7 (1.46) | -5.2 (1.53) | -5.4 (1.47)
  Presenteeism: number analyzed (Participants) | 173 | 145 | 166
  Presenteeism | -7.5 (2.49) | -22.2 (2.59) | -19.3 (2.46)
  Work productivity loss: number analyzed (Participants) | 173 | 145 | 166
  Work productivity loss | -7.2 (2.62) | -22.6 (2.73) | -20.2 (2.60)
  Activity impairment | -10.1 (2.07) | -24.7 (2.09) | -22.6 (2.04)

31. Secondary Outcome: Percentage of Participants With ≥5-Point Reduction From Baseline to Week 12 in HIT-6 Score
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 288 | 280 | 284
percentage of participants | 39.9 | 62.1 | 62.0

32. Secondary Outcome: Percentage of Participants With ≥5-Point Reduction From Baseline to Week 24 in HIT-6 Score
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 288 | 280 | 285
percentage of participants | 46.2 | 72.1 | 71.6

33. Secondary Outcome: Health Care Resource Utilization (HCRU): Visits to a Family Doctor/General Practitioner
Description: Number of participants who visited to a family doctor/general practitioner has been reported.
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 297 | 291 | 289
Participants
  0 Visit | 244 | 259 | 256
  1 Visit | 35 | 22 | 22
  2 Visits | 6 | 5 | 6
  3 Visits | 7 | 2 | 3
  4 Visits | 1 | 1 | 1
  5 Visits | 1 | 2 | 1
  6 Visits | 2 | 0 | 0
  8 Visits | 1 | 0 | 0

34. Secondary Outcome: HCRU: Visits to a Specialist
Description: Number of participants who visited to a specialist has been reported.
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 297 | 291 | 289
Participants
  0 Visit | 249 | 256 | 257
  1 Visit | 33 | 31 | 24
  2 Visits | 2 | 2 | 4
  3 Visits | 7 | 2 | 4
  5 Visits | 1 | 0 | 0
  6 Visits | 4 | 0 | 0
  8 Visits | 1 | 0 | 0

35. Secondary Outcome: HCRU: Number of Emergency Department Visits Due to Your Migraine
Description: Number of participants who visited to emergency department due to your migraine has been reported.
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 297 | 291 | 289
Participants
  0 Visit | 289 | 289 | 285
  1 Visit | 6 | 1 | 3
  2 Visits | 0 | 1 | 1
  3 Visits | 1 | 0 | 0
  8 Visits | 1 | 0 | 0

36. Secondary Outcome: HCRU: Number of Hospital Admissions Due to Migraine
Description: Number of participants who admitted in the hospital due to migraine has been reported.
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 297 | 291 | 289
Participants
  0 Visit | 295 | 289 | 287
  1 Visit | 1 | 1 | 2
  2 Visits | 0 | 1 | 0
  4 Visits | 1 | 0 | 0

37. Secondary Outcome: HCRU: Total Number of Overnight Hospital Stays Due to Migraine
Description: Number of participants who had total number of overnight hospital stays due to migraine has been reported.
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Eptinezumab 100 mg | Eptinezumab 300 mg
Number analyzed (Participants) | 297 | 291 | 289
Participants
  0 Visit | 295 | 290 | 289
  1 Visit | 1 | 0 | 0
  3 Visits | 1 | 1 | 0

38. Secondary Outcome: Change From Baseline in the Number of MMDs Averaged Over Weeks 25 to 36, 37 to 48, 49 to 60, and 61 to 72
Description: as for outcome 1
Time Frame: Baseline, Weeks 25 - 36, 37 - 48, 49 - 60, and 61 - 72
Population: Full-analysis-long-term set (FAS_LT) included all randomized participants who received at least 1 infusion of study drug, had a visit in the Extension Period, and who had a valid baseline assessment and a valid assessment of monthly migraine days in the Extension Period. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Error); unit: days/month
Groups:
- Placebo to Eptinezumab 100 mg: Participants who received placebo in the double-blind placebo-controlled period, received eptinezumab 100 mg in the dose-blinded extension period.
- Placebo to Eptinezumab 300 mg: Participants who received placebo in the double-blind placebo-controlled period, received eptinezumab 300 mg in the dose-blinded extension period.
- Eptinezumab 100 mg to Eptinezumab 100 mg: Participants who received eptinezumab 100 mg in the double-blind placebo-controlled period, continued to receive the same dose of eptinezumab in the dose-blinded extension period.
- Eptinezumab 300 mg to Eptinezumab 300 mg: Participants who received eptinezumab 300 mg in the double-blind placebo-controlled period, continued to receive the same dose of eptinezumab in the dose-blinded extension period.
Arm/Group | Placebo to Eptinezumab 100 mg | Placebo to Eptinezumab 300 mg | Eptinezumab 100 mg to Eptinezumab 100 mg | Eptinezumab 300 mg to Eptinezumab 300 mg
Number analyzed (Participants) | 144 | 146 | 282 | 282
days/month
  Change at Weeks 25-36 | -4.7 (0.49) | -6.1 (0.49) | -5.8 (0.39) | -5.9 (0.39)
  Change at Weeks 37-48: number analyzed (Participants) | 140 | 146 | 282 | 273
  Change at Weeks 37-48 | -5.0 (0.50) | -6.0 (0.50) | -5.8 (0.40) | -6.0 (0.40)
  Change at Weeks 49-60: number analyzed (Participants) | 134 | 140 | 270 | 265
  Change at Weeks 49-60 | -5.6 (0.51) | -6.6 (0.51) | -5.8 (0.41) | -6.0 (0.41)
  Change at Weeks 61-72: number analyzed (Participants) | 126 | 136 | 252 | 246
  Change at Weeks 61-72 | -5.9 (0.51) | -6.8 (0.51) | -6.6 (0.41) | -6.5 (0.41)

39. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in MMDs Averaged Over Weeks 25 to 36, 37 to 48, 49 to 60, and 61 to 72
Description: as for outcome 1
Time Frame: Baseline to Weeks 25 - 36, 37 - 48, 49 - 60, and 61 - 72
Population: FAS_LT included all randomized participants who received at least 1 infusion of study drug, had a visit in the Extension Period, and who had a valid baseline assessment and a valid assessment of monthly migraine days in the Extension Period. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Eptinezumab 100 mg | Placebo to Eptinezumab 300 mg | Eptinezumab 100 mg to Eptinezumab 100 mg | Eptinezumab 300 mg to Eptinezumab 300 mg
Number analyzed (Participants) | 144 | 146 | 282 | 282
percentage of participants
  Weeks 25-36 | 48.6 | 63.0 | 59.6 | 61.0
  Weeks 37-48: number analyzed (Participants) | 140 | 146 | 282 | 273
  Weeks 37-48 | 49.3 | 60.3 | 60.6 | 61.9
  Weeks 49-60: number analyzed (Participants) | 134 | 140 | 270 | 265
  Weeks 49-60 | 59.7 | 68.6 | 62.6 | 62.3
  Weeks 61-72: number analyzed (Participants) | 126 | 136 | 252 | 246
  Weeks 61-72 | 63.5 | 69.9 | 68.3 | 65.9

40. Secondary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in MMDs Averaged Over Weeks 25 to 36, 37 to 48, 49 to 60, and 61 to 72
Description: as for outcome 1
Time Frame: Baseline to Weeks 25 - 36, 37 - 48, 49 - 60, and 61 - 72
Population: as for outcome 39
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Eptinezumab 100 mg | Placebo to Eptinezumab 300 mg | Eptinezumab 100 mg to Eptinezumab 100 mg | Eptinezumab 300 mg to Eptinezumab 300 mg
Number analyzed (Participants) | 144 | 146 | 282 | 282
percentage of participants
  Weeks 25-36 | 19.4 | 28.1 | 25.9 | 31.2
  Weeks 37-48: number analyzed (Participants) | 140 | 146 | 282 | 273
  Weeks 37-48 | 27.9 | 30.8 | 31.6 | 32.6
  Weeks 49-60: number analyzed (Participants) | 134 | 140 | 270 | 265
  Weeks 49-60 | 32.1 | 33.6 | 29.3 | 38.9
  Weeks 61-72: number analyzed (Participants) | 126 | 136 | 252 | 246
  Weeks 61-72 | 36.5 | 39.0 | 37.7 | 44.7

41. Secondary Outcome: Change From Baseline in HIT-6 Score at Weeks 36, 48, 60, and 72
Description: as for outcome 5
Time Frame: Baseline, Weeks 36, 48, 60, and 72
Population: as for outcome 39
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo to Eptinezumab 100 mg | Placebo to Eptinezumab 300 mg | Eptinezumab 100 mg to Eptinezumab 100 mg | Eptinezumab 300 mg to Eptinezumab 300 mg
Number analyzed (Participants) | 138 | 139 | 265 | 272
units on a scale
  Change at Week 36: number analyzed (Participants) | 138 | 137 | 265 | 272
  Change at Week 36 | -10.01 (0.69) | -12.15 (0.73) | -10.99 (0.57) | -12.0 (0.56)
  Change at Week 48: number analyzed (Participants) | 134 | 139 | 260 | 260
  Change at Week 48 | -10.71 (0.77) | -12.71 (0.75) | -12.55 (0.59) | -12.68 (0.60)
  Change at Week 60: number analyzed (Participants) | 128 | 136 | 249 | 258
  Change at Week 60 | -12.54 (0.80) | -13.21 (0.71) | -12.57 (0.56) | -13.15 (0.59)
  Change at Week 72: number analyzed (Participants) | 124 | 131 | 239 | 237
  Change at Week 72 | -12.68 (0.87) | -15.02 (0.78) | -13.28 (0.63) | -14.13 (0.63)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72
Description: All-patients-treated set (APTS) included all randomized participants who received at least 1 infusion of the study drug. All-patients-treated-long-term set (APTS_LT) included all randomized participants who received at least 1 infusion of the study drug and had a visit in the Extension Period.
Groups:
- Placebo-controlled Period: Placebo: Participants received placebo matched to eptinezumab by IV infusion on Baseline (Day 0) and on Week 12.
- Placebo-controlled Period: Eptinezumab 100 mg; Placebo-controlled Period: Eptinezumab 300 mg: Participants received eptinezumab 100 mg by IV infusion on Baseline (Day 0) and on Week 12.
- Extension Period: Placebo to Eptinezumab 100 mg: Participants who received placebo in the double-blind placebo-controlled period, received eptinezumab 100 mg in the dose-blinded extension period.
- Extension Period: Placebo to Eptinezumab 300 mg: Participants who received placebo in the double-blind placebo-controlled period, received eptinezumab 300 mg in the dose-blinded extension period.
- Extension Period: Eptinezumab 100 mg to Eptinezumab 100 mg: Participants who received eptinezumab 100 mg in the double-blind placebo-controlled period, continued to receive the same dose of eptinezumab in the dose-blinded extension period.
- Extension Period: Eptinezumab 300 mg to Eptinezumab 300 mg: Participants who received eptinezumab 300 mg in the double-blind placebo-controlled period, continued to receive the same dose of eptinezumab in the dose-blinded extension period.
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Eptinezumab 100 mg | Placebo-controlled Period: Eptinezumab 300 mg | Extension Period: Placebo to Eptinezumab 100 mg | Extension Period: Placebo to Eptinezumab 300 mg | Extension Period: Eptinezumab 100 mg to Eptinezumab 100 mg | Extension Period: Eptinezumab 300 mg to Eptinezumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/299 | 0/294 | 0/145 | 0/148 | 0/288 | 0/284
Serious Adverse Events (participants affected / at risk) | 3/298 | 6/299 | 7/294 | 2/145 | 7/148 | 9/288 | 9/284
Other Adverse Events (participants affected / at risk) | 85/298 | 95/299 | 90/294 | 57/145 | 62/148 | 133/288 | 118/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-controlled Period: Placebo (N=298) | Placebo-controlled Period: Eptinezumab 100 mg (N=299) | Placebo-controlled Period: Eptinezumab 300 mg (N=294) | Extension Period: Placebo to Eptinezumab 100 mg (N=145) | Extension Period: Placebo to Eptinezumab 300 mg (N=148) | Extension Period: Eptinezumab 100 mg to Eptinezumab 100 mg (N=288) | Extension Period: Eptinezumab 300 mg to Eptinezumab 300 mg (N=284)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-controlled Period: Placebo (N=298) | Placebo-controlled Period: Eptinezumab 100 mg (N=299) | Placebo-controlled Period: Eptinezumab 300 mg (N=294) | Extension Period: Placebo to Eptinezumab 100 mg (N=145) | Extension Period: Placebo to Eptinezumab 300 mg (N=148) | Extension Period: Eptinezumab 100 mg to Eptinezumab 100 mg (N=288) | Extension Period: Eptinezumab 300 mg to Eptinezumab 300 mg (N=284)
Fatigue (General disorders) | 4 (4) | 2 (2) | 6 (6) | 0 (0) | 1 (1) | 5 (5) | 2 (3)
COVID-19 (Infections and infestations) | 16 (16) | 19 (19) | 15 (15) | 25 (26) | 31 (33) | 63 (69) | 63 (63)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (7) | 9 (11) | 7 (8) | 13 (15) | 19 (25) | 27 (38)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 5 (5) | 4 (5) | 1 (1) | 3 (4) | 4 (5) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (2) | 1 (1) | 1 (2) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (4) | 5 (5) | 1 (2) | 5 (5) | 2 (2) | 3 (3)
Asthenia (General disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 4 (4) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 5 (6)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 4 (4) | 6 (8) | 13 (14) | 8 (8)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (1) | 5 (5) | 3 (4) | 4 (4) | 3 (4) | 4 (5)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Blood pressure increased (Investigations) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 4 (5) | 1 (1) | 2 (3) | 6 (6) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 3 (3) | 1 (1) | 2 (2) | 8 (8) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 2 (3) | 4 (5)
Headache (Nervous system disorders) | 3 (4) | 3 (4) | 3 (3) | 2 (3) | 2 (3) | 3 (3) | 1 (1)
Migraine (Nervous system disorders) | 3 (3) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 7 (7) | 2 (4)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 3 (3) | 4 (4) | 4 (4) | 3 (4) | 0 (0) | 3 (4) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
Haemorrhoids (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Immunisation reaction (Immune system disorders) | 2 (3) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 3 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 4 (5)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Weight increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Menopause (Social circumstances) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT04418765/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT04418765/SAP_001.pdf